CLINICAL TRIAL: NCT05758376
Title: Recovery Bridge: A Peer Facilitated Intervention to Help Bridge the Transition From Psychiatric Inpatient Hospitalized to Living in the Community
Brief Title: Recovery Bridge: Peer Intervention to Bridge Transition Post Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 22-004
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mental Illness
Keywords: Veteran; In-patient
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Open Pilot Trial (n=15) to examine feasibility, fidelity, and acceptability of study intervention (called Recovery Bridge)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Recovery Bridge (Experimental): Open trial single arm pilot study
  Interventions: Behavioral: Recovery Bridge

INTERVENTIONS:
Behavioral: Recovery Bridge — Recovery Bridge is a Peer Specialist facilitated intervention designed to help Veterans being discharged from an inpatient psychiatric hospitalization bridge the gap to outpatient care and community living

SUMMARY:
The time following discharge from psychiatric hospitalization is a high-risk period and has been associated with a range of negative outcomes including high rates of hospital readmission and suicide. The purpose of this proposal is to: 1) create a Peer Specialist facilitated intervention, called Recovery Bridge, designed to facilitate the transition from inpatient psychiatric hospitalization to community living; 2) examine feasibility, fidelity, and acceptability; and preliminarily explore the impact of the intervention on: a) readmission rates and connection to outpatient care compared to a control group identified from administrative data; and b) change in recovery and quality of life measures over time in the intervention participants. Results from the proposed open pilot trial will set the stage for next steps including a larger effectiveness trial followed by a possible hybrid-I effectiveness/implementation trial to inform future dissemination and implementation of the intervention more broadly across the VA.

DETAILED DESCRIPTION:
Background: The time following discharge from psychiatric hospitalization is a high-risk period and has been associated with a range of negative outcomes, including high rates of hospital readmission and suicide (1). Because the evidence for transitional discharge interventions with bridging components is mixed and limited in terms of how Peer Specialists (PS) can help support such interventions, additional research is needed. This proposal calls for the development and preliminary evaluation of a PS facilitated technology-supported intervention based on the existing and frequently used My Recovery Plan program. However, to date, no studies have examined use of this tool to improve post-hospital discharge outcomes. Given the importance of the problem for the VA, and the fact that the VA has both a large PS infrastructure that is valued by both professional providers and Veterans, the investigators' work offers sound justification and the unique opportunity to test the proposed intervention in a single integrated system of inpatient and outpatient services.

Significance: The significance of this project lies in its ability to actively address an important gap in the research, namely PS interventions focused on reducing readmission and supporting recovery-oriented outcomes in Veterans. Further relating to important HSR&D priorities the project is designed to advance scientific knowledge and clinical practice in the areas of access to care, mental health, and suicide prevention.

Innovation and Impact: A key innovation of the proposed research is the potential to efficiently optimize existing resources to target the widespread challenges associated with transitioning out of acute inpatient settings and effectively connect Veterans to preferred services (in this case peer support) in order to prevent re-admission, and improve utilization of VA outpatient mental health services. Finally, in relationship to impact, Recovery Bridge has potential to result in improvement across multiple clinical and functional outcomes that are applicable to a broad Veteran population (rather than only in small select diagnostically specific subpopulations).

Specific Aim 1: Integrate the My Recovery Plan tool and existing PS tools and strategies to develop a manualized intervention called Recovery Bridge for use by VA PS working to help Veterans make the transition from acute inpatient psychiatric hospitalization to community living.

Specific Aim 2: Complete an open pilot trial (n=15) to examine the feasibility, fidelity, and acceptability of the Recovery Bridge intervention in relation to well specified benchmarks supporting continued and expanded investigation.

[Specific Aim 3: As part of the open pilot trial: 1) explore the impact of the intervention on readmission rates (at 30 and 90 days), and connection to outpatient care compared to a control group (n=15) identified from administrative data, and; 2) explore the change in recovery and Quality of Life measures over time in the intervention participants].

Methodology: Source documents described in the proposal will be used to create the Recovery Bridge intervention (as Specified in Aim 1). Quantitative, qualitative, and administrative services data the investigators will be used to complete an open trial of the intervention (as specified in Aim 2 and Aim 3).

Next Steps: Benchmarks across the domains of feasibility, fidelity, and acceptability; as well as exploratory outcomes specified in Aim 3, will be used to inform next steps including a larger effectiveness trial followed by a possible hybrid-I effectiveness/implementation trial to inform future dissemination and implementation of the intervention more broadly across the VA.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for active sample:

* 18 years of age or older
* enrolled in the inpatient program
* planned discharge to the community

Exclusion Criteria:

* Inability to provide consent
* No access to either a computer or a telephone after discharge (as at least one of these will be needed should the Veteran and PS interventionist decide to continue to meet remotely)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Goldberg, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single Arm Open Trial (for primary outcomes)
  The primary outcomes in this open trial were only for the single arm actively recruited for the study
Period: Overall Study
Arm/Group | Recovery Bridge
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recovery Bridge
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 4
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility 1: Recruitment Benchmark
Description: Recruitment (number consented divided by number approached)
Time Frame: 3 months
Population: Overall Number of Participants Analyzed reflects the number of participants approached
Measure: Number; unit: participants
Arm/Group | Recovery Bridge
Number analyzed (Participants) | 27
participants | 15

2. Primary Outcome: Feasibility 2: Intervention Engagement (Percentage of Sample That Completes at Least 3 Intervention Sessions-with One of the Three Occurring Inpatient
Description: Percentage of sample that completes at least 3 intervention sessions-with one of the three occurring inpatient
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Recovery Bridge
Number analyzed (Participants) | 15
Participants | 13

3. Primary Outcome: Feasibility 3: Drop Out Rate (Percent That Did Not Complete Post-intervention Assessment)
Description: Drop out Rate: Percent that do not complete post-intervention assessment (based on count of participants)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Recovery Bridge
Number analyzed (Participants) | 15
Participants | 5

4. Primary Outcome: Fidelity
Description: Greater than 90% of all Adherence and Competence Items Rated as Acceptable or Higher. Higher ratings of acceptability are considered to be the better outcome.
Time Frame: 3 months
Population: among the sessions reviewed for fidelity across the two criteria (adherence and competence)
Measure: Number; unit: % of reviewed sessions meeting fidelity
Units Other Than Participants: number-of-recorded-sessions
Arm/Group | Recovery Bridge
Number analyzed (Participants) | 15
Number analyzed (number-of-recorded-sessions) | 15
% of reviewed sessions meeting fidelity | 93

5. Primary Outcome: Acceptability (Patient Satisfaction Questionnaire--administered Post Intervention)
Description: Score of 26 percent or higher on Patient Satisfaction Questionnaire. Scale ranges from 8-32, higher score is associated with "better outcome" (i.e. higher satisfaction).
Time Frame: 3 months
Population: only those completing intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovery Bridge
Number analyzed (Participants) | 10
score on a scale | 27.1 (4.2)

ADVERSE EVENTS:
Time Frame: from baseline until post-assessment (up to 3 months)
Arm/Group | Recovery Bridge
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT05758376/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT05758376/ICF_000.pdf